CLINICAL TRIAL: NCT06007547
Title: Prophylactic Minimally Invasive Surfactant Evaluation
Acronym: PreProMISe
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Endeavor Health (Other)
Collaborators: Chiesi USA, Inc. (Industry)
Responsible Party: Principal Investigator, Matthew Derrick, Attending Neonatologist, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EH23-107
Record Dates: First submitted 2023-07-27; First posted 2023-08-23 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Respiratory Distress Syndrome, Newborn; Premature Birth
Keywords: Respiratory Distress Syndrome; surfactant; Minimally invasive Surfactant Therapy
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Premature Birth; Respiratory Distress Syndrome | interventions — poractant alfa

STUDY DESIGN:
Intervention Model Description: Comparison of prophylaxis compared to rescue surfactant, administered using a minimally invasive technique, in premature infants less that 30 weeks gestation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Prophylactic Surfactant via Minimally Invasive Technique (Experimental): Infants randomized to prophylactic surfactant treatment will receive a dose of poractant alfa (Curosurf) administered under direct laryngoscopy using a surfactant instillation catheter (MIST) 16G Angiocath (Becton Dickinson, Sandy, UT, USA), at a dosage of 200 mg/kg as soon as possible after delivery (within 15 minutes).
  Interventions: Drug: Poractant Alfa
- Rescue Surfactant via Minimally Invasive Technique (Active Comparator): The control group will be given surfactant will receive a dose of poractant alfa (Curosurf) administered under direct laryngoscopy using a surfactant instillation catheter (MIST) 16G Angiocath (Becton Dickinson, Sandy, UT, USA), at a dosage of 200 mg/kg if their fiO2 reaches a threshold of ≥30% within the first 48 hours of life.
  Interventions: Drug: Poractant Alfa

INTERVENTIONS:
Drug: Poractant Alfa — Poractant alfa (Curosurf) 200mg/kg administered under direct laryngoscopy using a surfactant instillation catheter
  Other Names: Minimally Invasive Surfactant Therapy

SUMMARY:
The purpose of this study is to explore the question: Does prophylactic administration of exogenous surfactant in the delivery room, using a minimally-invasive technique, improve outcome in preterm infants 22-29 weeks' gestation compared to rescue treatment using the same technique?

DETAILED DESCRIPTION:
RESEARCH DESIGN Multicenter, randomized, controlled trial.

Northshore Evanston Hospital will be the primary site. It is hoped that Northwest Community, University of Chicago, Edwards Hospital, Advocate Park Ridge, Advocate Oak Lawn and Advocate Illinois Masonic will also join the study.

RECRUITMENT Entry criteria Inborn preterm infants 22 0/7-29 6/7 weeks' gestation, with be randomized to prophylactic Minimally Invasive Surfactant Therapy (MIST) in the delivery room compared to rescue MIST if fraction of inspired oxygen (FiO2) ≥0.30 at less than 48 hours of age. Babies in both groups will be managed on nasal continuous positive airway pressure (NCPAP) pressures of 5-8 cm water.

Exclusion criteria Infants will be excluded if there is a congenital anomaly or an alternative cause for respiratory distress.

Babies who require emergent intubation in the delivery room will not be enrolled in the interventions.

Parental Consent will be obtained prior to birth. Once delivery is imminent infant will be randomized to immediate versus rescue surfactant administration via MIST. Randomization will be in blocks of 6 and using cards with created by a web based randomizer.

Infants who require emergent intubation in the delivery room will not be enrolled in the interventions but their clinical outcomes will be assessed the same as the babies who receive the intervention.

There will be three gestational age strata (22-23 weeks, 24-26 weeks and 27-29 weeks). Twins and higher order multiples will be randomized independently. Babies in the lowest gestational age strata will not be enrolled at a center until 5 babies at that center have been enrolled in either of the other groups.

INTERVENTION Infants randomized to prophylactic surfactant treatment will receive a dose of poractant alfa (Curosurf) administered under direct laryngoscopy using a surfactant instillation catheter (MIST) 16 Gauge Angiocath (Becton Dickinson, Sandy, UT, USA), at a dosage of 200 mg/kg as soon as possible after delivery (within 15 minutes). The infants will be stabilized and placed on NCPAP or High flow Nasal Cannula (HFNC).

Briefly the MIST procedure is as follows: the angiocath is inserted to an appropriate depth under direct laryngoscopy, the laryngoscope is removed, a carbon dioxide (CO2) detector is placed on the end of the catheter with a endotracheal tube adaptor. If the color changes then adaptor and detector are removed and the surfactant is instilled over about 1 minute and the catheter is removed. The infant is maintained on NCPAP/HFNC during the procedure.

Infants of both groups will be supported via HFNC or NCPAP in the delivery room and then transitioned to NCPAP in the neonatal intensive care unit (NICU).

The control group will be given surfactant via MIST if their fiO2 reaches a threshold of ≥30% within the first 48 hours of life.

A second dose of poractant alfa (Curosurf), at a dosage of 100mg/kg, will be administered via MIST to both groups if their fiO2 reaches the threshold of 30% between 6 and 48 hours after the first dose.

No further surfactant should be given in the first 7 days unless the infant reaches the intubation criteria.

POST-INTERVENTION MANAGEMENT Other than the requirement to adhere to intubation criteria in the first week, and in some cases perform a room air trial at 36 weeks corrected gestation, management will be at the discretion of the clinical team.

Titration of CPAP pressure is encouraged, with a permitted maximum of 8 cm H2O. Use of nasal intermittent positive-pressure ventilation (NIPPV) is allowable for apnea, but discouraged for Respiratory Distress Syndrome (RDS) and should only be after at least one dose of surfactant has been given.

Early caffeine therapy is expected.

Criteria for intubation:

Enrolled infants on CPAP will be intubated if:

* FiO2 ≥0.45 for 15 minutes, or if there is unremitting apnea (> 6 episodes/hour requiring intervention or in the opinion of the treating physician) or persistent respiratory acidosis (pH<7.25 and partial pressure of carbon dioxide (pCO2) >60) on blood gasses at least 30 minutes apart or metabolic acidosis refractory to treatment.
* Need for an anesthetic or an intervention requiring intubation

These criteria apply during the first week of life, and to the first episode of intubation only. If the infant is intubated it is expected that another dose of surfactant will be administered.

OUTCOMES Primary outcome: Intubation in the first 7 days of age.

Secondary outcomes:

* Respiratory Incidence of composite outcome of death or physiological bronchopulmonary dysplasia (BPD). Durations of mechanical respiratory support, CPAP, high flow nasal cannula, (HFNC), oxygen therapy. Pneumothorax or pulmonary hemorrhage.
* Non respiratory neonatal morbidities intraventricular hemorrhage, periventricular leukomalacia, retinopathy of prematurity, necrotizing enterocolitis, and patent ductus arteriosus. Corrected age at discharge, length of hospital stay (a proxy for cost). Neonatal follow up data.

The above data will be collected until discharge. Babies born between 22 and 29 weeks are routinely followed by our developmental follow up clinic. The information from the 2-year developmental clinic visit will be recorded by the study.

SAMPLE SIZE 200, 50 being from NorthShore. Between 2018 and 2022 65% of the babies in this gestational age had an endotracheal tube inserted at Evanston Hospital, and were ventilated. Detection of a reduction of 25% (from 65% to 40%) with a 90% power and α = 0.05 (two-sided) would require 82 subjects per arm. It is anticipated that patient recruitment should take 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age <30 weeks
* Antenatal consent from Parent

Exclusion Criteria:

* Congenital anomalies
* Alternate cause of respiratory distress

Max Age: 15 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Endotracheal Intubation | 7 days
  Oxygen requirement > 45% requiring endotracheal intubation

SECONDARY OUTCOMES:
Bronchopulmonary dysplasia | 36 weeks corrected gestational age
  Oxygen requirement to 36 weeks corrected age

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Derrick, MBBS, Principal Investigator — Northshore Univ Healthsystem
Locations (1):
- Northshore University Healthsystem, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dargaville PA, Kamlin COF, Orsini F, Wang X, De Paoli AG, Kanmaz Kutman HG, Cetinkaya M, Kornhauser-Cerar L, Derrick M, Ozkan H, Hulzebos CV, Schmolzer GM, Aiyappan A, Lemyre B, Kuo S, Rajadurai VS, O'Shea J, Biniwale M, Ramanathan R, Kushnir A, Bader D, Thomas MR, Chakraborty M, Buksh MJ, Bhatia R, Sullivan CL, Shinwell ES, Dyson A, Barker DP, Kugelman A, Donovan TJ, Tauscher MK, Murthy V, Ali SKM, Yossuck P, Clark HW, Soll RF, Carlin JB, Davis PG; OPTIMIST-A Trial Investigators. Effect of Minimally Invasive Surfactant Therapy vs Sham Treatment on Death or Bronchopulmonary Dysplasia in Preterm Infants With Respiratory Distress Syndrome: The OPTIMIST-A Randomized Clinical Trial. JAMA. 2021 Dec 28;326(24):2478-2487. doi: 10.1001/jama.2021.21892. PMID 34902013
- [Background] Kendig JW, Notter RH, Cox C, Reubens LJ, Davis JM, Maniscalco WM, Sinkin RA, Bartoletti A, Dweck HS, Horgan MJ, et al. A comparison of surfactant as immediate prophylaxis and as rescue therapy in newborns of less than 30 weeks' gestation. N Engl J Med. 1991 Mar 28;324(13):865-71. doi: 10.1056/NEJM199103283241301. PMID 2000109
- [Background] Kribs A, Hartel C, Kattner E, Vochem M, Kuster H, Moller J, Muller D, Segerer H, Wieg C, Gebauer C, Nikischin W, Wense Av, Herting E, Roth B, Gopel W. Surfactant without intubation in preterm infants with respiratory distress: first multi-center data. Klin Padiatr. 2010 Jan-Feb;222(1):13-7. doi: 10.1055/s-0029-1241867. Epub 2010 Jan 18. PMID 20084586
- [Background] Kattwinkel J, Bloom BT, Delmore P, Davis CL, Farrell E, Friss H, Jung AL, King K, Mueller D. Prophylactic administration of calf lung surfactant extract is more effective than early treatment of respiratory distress syndrome in neonates of 29 through 32 weeks' gestation. Pediatrics. 1993 Jul;92(1):90-8. PMID 8516091
- [Background] SUPPORT Study Group of the Eunice Kennedy Shriver NICHD Neonatal Research Network; Finer NN, Carlo WA, Walsh MC, Rich W, Gantz MG, Laptook AR, Yoder BA, Faix RG, Das A, Poole WK, Donovan EF, Newman NS, Ambalavanan N, Frantz ID 3rd, Buchter S, Sanchez PJ, Kennedy KA, Laroia N, Poindexter BB, Cotten CM, Van Meurs KP, Duara S, Narendran V, Sood BG, O'Shea TM, Bell EF, Bhandari V, Watterberg KL, Higgins RD. Early CPAP versus surfactant in extremely preterm infants. N Engl J Med. 2010 May 27;362(21):1970-9. doi: 10.1056/NEJMoa0911783. Epub 2010 May 16. PMID 20472939